CLINICAL TRIAL: NCT06703554
Title: The Impact of Natural Sage Extract on Glucosyltransferase B and D Gene Expression in Streptococcus Mutans: A Randomized Clinical Trial Using Real Time Polymerase Chain Reaction
Brief Title: The Impact of Sage Extract on GTS B and D Gene Expression in S. Mutans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Ezz, Lecturer at Conservative Department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Sage Extract
Record Dates: First submitted 2024-11-10; First posted 2024-11-25 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Caries,Dental; Dental Caries; Dental Diseases
Keywords: High caries risk; Chlorohexidine; Real-time PCR
MeSH Terms: conditions — Dental Caries; Stomatognathic Diseases | interventions — Biological Products

STUDY DESIGN:
Intervention Model Description: Sage Extract Natural product
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: same bottles dark in color was used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sage oil mouthwash (Experimental): Sage oil obtained from a local market of herbal products in Egypt. In order to identify chemical composition of sage essential oils and overall purity, Gas Chromatography/ Mass Spectrometry analysis (GC/MS) performed
  Interventions: Other: Sage Oil Mouthwash
- Chlorohexidine Mouthwash (Active Comparator): 0.12% chlorhexidine gluconate in a base containing water, 11.6% alcohol, glycerin, PEG-40 sorbitan diisostearate, flavor, and sodium saccharin
  Interventions: Biological: Chlorohexidine Mouthwash

INTERVENTIONS:
Other: Sage Oil Mouthwash — Sage oil obtained from a local market of herbal products in Egypt. In order to identify chemical composition of sage essential oils and overall purity, Gas Chromatography/ Mass Spectrometry analysis (GC/MS) performed
  Other Names: Natural product
  Arms: Sage oil mouthwash
Biological: Chlorohexidine Mouthwash — 0.12% chlorhexidine gluconate in a base containing water, 11.6% alcohol, glycerin, PEG-40 sorbitan diisostearate, flavor, and sodium saccharin
  Other Names: CHX mouthwash
  Arms: Chlorohexidine Mouthwash

SUMMARY:
Glucosyltransferases (Gtfs) play a crucial role in the pathogenesis of dental caries caused by Streptococcus mutans. Gtfs is recognized as an attractive target for effective therapeutic interventions aimed at inhibiting cariogenic biofilms.

Objective: This study evaluates the antibacterial effects of sage extract compared to chlorhexidine mouthwashes on the expression of Gtf genes in S. mutans from salivary samples of high caries risk patients over a one-month follow-up, utilizing real-time polymerase chain reaction.

Methodology: This clinical trial involves 42 participants with a high risk for caries, who are randomly divided into two groups of 21 subjects each.

DETAILED DESCRIPTION:
Glucosyltransferases (Gtfs) are essential in the development of dental caries caused by Streptococcus mutans. They are currently recognized as promising targets for effective therapeutic strategies aimed at disrupting cariogenic biofilms.

Objective: This study investigates the antibacterial effects of sage extract in comparison to chlorhexidine mouthwashes on the expression of Gtf genes in S. mutans from the saliva of patients at high risk for caries, over a one-month follow-up period, using real-time polymerase chain reaction.

Methodology: This clinical trial includes 42 high caries risk participants, who are randomly assigned to two groups, each consisting of 21 subjects.

ELIGIBILITY:
Inclusion Criteria:

* medically free, high caries patient with DMFT

Exclusion Criteria:

* pregnant and smokers

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
real-time PCR | 1 week
  S. Mutans, Gtf B, Gtf D
real-time PCR | 2 weeks
  S. Mutans, Gtf B, Gtf D
real-time PCR | 3 weeks
  S. Mutans, Gtf B, Gtf D
real-time PCR | 4 weeks
  S. Mutans, Gtf B, Gtf D
Gene Expression | 1 week
  S. Mutans, Gene Expression
Gene Expression | 2 weeks
  S. Mutans, Gene Expression
Gene Expression | 3 weeks
  S. Mutans, Gene Expression
Gene Expression | 4 weeks
  S. Mutans, Gene Expression

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No